CLINICAL TRIAL: NCT01990287
Title: SENSE (Subcutaneous and Epidural Neuromodulation System Evaluation)Study for the Treatment of Chronic Low Back and Leg Pain
Brief Title: SENSE (Subcutaneous and Epidural Neuromodulation System Evaluation) Study
Acronym: SENSE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-11-12
Record Dates: First submitted 2013-11-15; First posted 2013-11-21 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Failed Back Surgery Syndrome; Post-Laminectomy Syndrome; Low Back Pain
Keywords: Low Back Pain; Failed Back surgery Syndrome; Post-Laminectomy Syndrome; Spinal Cord Stimulation; Peripheral Nerve field Stimulation; Pain
MeSH Terms: conditions — Failed Back Surgery Syndrome; post laminectomy syndrome; Low Back Pain; Pain | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SCS and PNfS (Experimental): Eon or Eon Mini IPG with epidural leads in the spinal column and subcutaneous leads in the peripheral field
  Interventions: Device: SCS and PNfS
- SCS Alone (Active Comparator): Eon or Eon Mini IPG with epidural leads in the spinal column
  Interventions: Device: SCS Alone

INTERVENTIONS:
Device: SCS and PNfS — Spinal Cord Stimulation (SCS) in combination with Peripheral Nerve Field Stimulation (PNfS). The SCS leads will be placed in the Thoracolumbar region and the PNfS lead will be placed subcutaneously in the area of pain.
  Other Names: Eon or Eon Mini IPG neurostimulation system with associated components
  Arms: SCS and PNfS
Device: SCS Alone — Spinal Cord Stimulation (SCS) only. The SCS leads will be placed in the Thoracolumbar region only.
  Other Names: Eon or Eon Mini IPG neurostimulation system with associated components
  Arms: SCS Alone

SUMMARY:
The purpose of the study is to demonstrate safety and efficacy of spinal cord stimulation with peripheral nerve field stimulation for the treatment of chronic low back and leg pain.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject is 22 years of age or older
* Subject has chronic low back and leg pain secondary to Failed Back Surgery Syndrome (FBSS)
* Subject has an average score of 6 or higher for average daily overall pain on the Numerical Rating Scale (NRS) based on the 7 day pain diary
* Subject has attempted "best" medical therapy and has tried and failed at least three documented medically supervised treatments (including, but not limited to physical therapy, acupuncture, etc.) and has failed medication treatment from at least two different classes
* Subject's pain-related medication regimen is stable 4 weeks prior to the baseline evaluation
* Subject agrees not to add or increase pain-related medication throughout the 12 week randomized evaluation phase of the study (starting at activation)

Key Exclusion Criteria:

* Subject currently participating in a clinical investigation that includes an active treatment arm
* Subject has been implanted with a previous neuromodulation system (PNfS, SCS-PNfS or SCS) or participated in a trial for a neuromodulation system
* Subject's overall Beck Depression Inventory II Score is > 24 or has a score of 3 on question 9 relating to suicidal thoughts or wishes at the baseline visit
* Subject with an infusion pump or any implantable neurostimulator device
* Subject has an existing medical condition that is likely to require repetitive MRI evaluation in the future (i.e. epilepsy, stroke, multiple sclerosis, acoustic neuroma, tumor)
* Subject has an existing medical condition that is likely to require the use of diathermy in the future
* Subject has peripheral vascular disease
* Subject is immunocompromised
* Subject has documented history of allergic response to titanium or silicone
* Subject has a documented history of substance abuse (narcotics, alcohol, etc.) or substance dependency in the 6 months prior to baseline data collection
* Female candidates of child bearing potential that are pregnant (confirmed by positive pregnancy test)

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-11; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Safety | 6 months
  Evaluation of device or procedure related adverse events
Efficacy | 3 months
  Responder rate in SCS-PNfS vs SCS alone

SECONDARY OUTCOMES:
Quality of Life | 3 months
Functional Disability | 3 months
Worst pain | 3 months
Rescue medication usage | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Porter McRoberts, MD, Principal Investigator — Holy Cross Orthopedic Institute
Locations (28):
- United States (28):
  - The Pain Center of Arizona, Phoenix, Arizona
  - Valley Pain Consultants - N. Scottsdale, Scottsdale, Arizona
  - Arizona Pain Specialists, Scottsdale, Arizona
  - The Mocek Spine Clinic, Little Rock, Arkansas
  - Comprehensive Pain Management Center, Campbell, California
  - Coastal Pain & Spinal Diagnostics Medical Group, Carlsbad, California
  - Pacific Pain Medicine Consultants, Oceanside, California
  - Pasadena Rehabilitation Institute, Pasadena, California
  - Bright Health Physicians of PIH, Whittier, California
  - Comprehensive Pain Specialists, Broomfield, Colorado
  - Holy Cross Orthopedics, Fort Lauderdale, Florida
  - H. Lee Moffitt Cancer and Research Institute, Tampa, Florida
  - Pain Care LLC, Stockbridge, Georgia
  - Interventional Pain Care, Muncie, Indiana
  - Bluegrass Pain, Louisville, Kentucky
  - Mid Atlantic Spine and Pain Physicians, Elkton, Maryland
  - Michigan Pain Specialists, Brighton, Michigan
  - Comprehensive Pain & Rehabilitation, Pascagoula, Mississippi
  - Neurological Surgery, P.C., Lake Success, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Carolina Pain Institute, Winston-Salem, North Carolina
  - Integrated Pain Solutions, Columbus, Ohio
  - Pain and Spine Center, Dayton, Ohio
  - Performance Spine and Sports Physicians, P.C., Pottstown, Pennsylvania
  - Vertex Spine and Pain, Franklin, Tennessee
  - Granger Pain and Spine, West Jordan, Utah
  - The Center for Pain Relief, Charleston, West Virginia